CLINICAL TRIAL: NCT03242525
Title: Examination of the Time Advantage of Point of Care Testing (POCT) Compared to the Conventional Central Laboratory Analysis in Intraclinical Patient Care
Brief Title: Examination of the Time Advantage Between POCT and Conventional Central Laboratory Analysis
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Florian Raimann, Dr. med., Johann Wolfgang Goethe University Hospital
Other Study IDs: 279/17
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Blood; Point-of-Care Systems; Analysis, Event History

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergency room: Twelve bleeding patients who are assigned to the emergency department receive a simultaneous blood analysis with POCT and central laboratory.
  Interventions: Diagnostic Test: POCT and central laboratory blood analysis
- Delivery room: Twelve bleeding patients who are assigned to the delivery room receive a simultaneous blood analysis with POCT and central laboratory.
  Interventions: Diagnostic Test: POCT and central laboratory blood analysis

INTERVENTIONS:
Diagnostic Test: POCT and central laboratory blood analysis — In every participant blood analysis will be performed by POCT and central laboratory investigating the time advantage.

SUMMARY:
The aim of the present study is to quantify the time advantage achieved by the use of POCT compared to conventional coagulation diagnostics. A further objective of this study is an analysis of the result quality of POCT for the prothrombin time / international normalized ratio.

DETAILED DESCRIPTION:
In order to be able to carry out a targeted coagulation therapy for the time-critical treatment of coagulopathic emergency patients, knowledge of the hemostatic potential is necessary.

After taking blood samples for coagulation diagnostics, they are sent to the central laboratory. After the analysis and validation the electronic provision of the results takes place. The loss of time by sample transport, analysis and breadth of the results extends the duration until therapy can be started.

The period of time until these analysis results are determined depends on several factors like daytime, day of week and location of the sample consignor and the availability of the laboratory. Not every clinic is connected to an internal tube mail system so that the samples have to be sent partly with a transport service.

In recent years, Point of Care (POCT) devices have become an increasingly important tool for diagnosing coagulopathic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years

Exclusion Criteria:

* Missing written consent
* Withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All bleeding patients assigned to the emergency department and delivery room.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Time advantage | 2-4 hours
  Duration until laboratory results are available after sampling for central laboratory versus POCT

SECONDARY OUTCOMES:
Correlation between central laboratory and POCT results. | 2-4 hours
  Correlation of prothrombin time / international normalized ratio results between POCT and central laboratory analysis.
Influence of transport type. | 2-4 hours
  Difference of results availability weather probes are transported by transport service or tube-mail.
Influence of daytime and weekday on results availability. | 2-4 hours
  Difference of results availability in dependence of daytime and weekday on transport duration.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zacharowski, Prof. Dr., Study Director — Department of Anesthesia, Intensive Care Medicine and Pain Therapy
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No